CLINICAL TRIAL: NCT05042232
Title: Assessing Behavioral, Functional, and Clinical Patient-Reported Outcomes (PROs) in Subjects Diagnosed With COVID-19
Brief Title: A Prospective Virtual Study of Patient Reported Behaviors and Health Outcomes in Individuals With COVID-19
Status: Completed | Type: Observational
Sponsor: Everly Health (Industry)
Responsible Party: Sponsor
Other Study IDs: EW-US-4010-0003
Record Dates: First submitted 2021-09-09; First posted 2021-09-13 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Other: SARS-CoV-2 Positive — Participants who have tested positive for SARS-CoV-2, both with and without symptoms
Other: SARS-CoV-2 Negative — Participants who have tested negative for SARS-CoV-2

SUMMARY:
The primary objective of this study is to identify and describe patient behaviors and clinical outcomes among patients who have tested positive for mild to moderate COVID-19.

DETAILED DESCRIPTION:
This virtual observational cohort study will describe patient behaviors and clinical outcomes of subjects who tested positive for COVID-19. Among those with positive tests, predictors of time to recovery, post-COVID function and outcomes will be identified. Individuals who test negative and positive for SARS-CoV-2 will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Individuals with a valid diagnostic COVID-19 test result

Exclusion Criteria:

- Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who have valid COVID-19 test results.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
To identify and describe patient behaviors and clinical outcomes among patients who have tested positive for COVID-19 | Up to 12 months

SECONDARY OUTCOMES:
To describe recovery in patients with test-confirmed COVID-19 infection including time to recovery and functional improvement | Up to 12 months
To develop prediction tools for time to recovery, function and outcomes in patients with COVID-19 identified by home testing | Up to 12 months
To describe users and the utilization of COVID-19 home testing over time by geography, demographics, and comorbidity | Up to 12 months
To describe the feasibility of COVID-19 home testing | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bauer, PhD, Principal Investigator — Everly Health
Locations (1):
- Everlywell, Inc, Austin, Texas, United States